CLINICAL TRIAL: NCT03677245
Title: The Effect of Balance Bike Training on Balance, Physical Activity Levels, and Participation in Children and Youth Down Down Syndrome: a Pilot Study
Brief Title: Balance Bike Training in Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0070
Record Dates: First submitted 2018-09-11; First posted 2018-09-19 (Actual); Results first posted 2020-04-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Down Syndrome; Postural Balance
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Intervention Model Description: pre- post-test design with each participant serving as his or her own control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Balance Biking (Experimental): Strider Balance Bike riding for 5 days following the Strider Learn to Ride Curriculum
  Interventions: Other: Strider Balance Bike

INTERVENTIONS:
Other: Strider Balance Bike — Learning to ride a Strider balance bike

SUMMARY:
Background: Children with Down syndrome (DS) present with hypotonia, impaired balance and poor gross motor proficiency which lead to difficulty learning new motor skills, decreased engagement in physical activity, and limited participation in home, school, and community activities. Bicycle riding is a popular childhood activity with multiple health benefits; however, children with DS often have difficulty learning to ride a standard two-wheel bike. Purpose: The purpose of this pilot study is to determine the effectiveness of the Strider "Learn to Ride" intervention when used to teach children with DS to ride a two-wheel balance bike. Additional purposes include examining the immediate effects of the five-day "Learn to Ride" intervention on the balance of children with DS and the long-term effects of completion of the intervention on the participation and physical activity levels of children with DS. Methods: An estimated 10 children between the ages of 5 and 17 years old will be recruited to participate in this pre- post-test group design study. The participants will complete the five-day Strider "Learn to Ride" intervention under the instruction of a pediatric physical therapist. The immediate effects of the intervention on distance cycled and balance, using the Pediatric Balance Scale (PBS), will be assessed. Participation and physical activity levels will be assessed at long term follow-up using the Participation and Environment Measure for Children and Youth (PEM-CY) and a PROMIS physical activity questionnaire.

DETAILED DESCRIPTION:
The proposed pilot study is a pre- post-test design with each participant serving as his or her own control. Children and adolescents with Down syndrome will be recruited from pediatric physical therapy clinics, local school districts, and the Central Mississippi Down Syndrome Association. Flyers will be provided to local pediatric therapy clinics and school districts. The director of the Central Mississippi Down Syndrome Association will be contacted by the PI (see email attached) and asked to send out a target recruitment email to all families of children with Down syndrome that are on the Central Mississippi Down Syndrome Association email list. To be included in the study, the individuals must 1) be between the ages of 5 and 17 years old with a diagnosis of Down syndrome, 2) have the core strength and balance necessary to maintain sitting on a two-wheel bike with their feet on the ground, and 3) be able to follow simple commands. The exclusion criteria for the study are 1) significant cardiovascular event or illness in the past 6 months and 2) another medical diagnosis, besides Down syndrome, that would limit participation in the exercise programs. The Institutional Review Board at the University of Mississippi Medical Center will approve all procedures. Each participant will complete an assent form to participate. Each participant will complete an assent and each parent/caregiver will complete an informed consent prior to enrolling their child in the study. If the child is unable to provide assent, due to age and/or cognitive deficits, only parental permission will be obtained. Additionally, each participant's parent/caregiver will be asked to complete the "registration packet" (attached to the IRB) in order to provide the researchers with health-related information that may be needed to ensure participant safety during the intervention sessions. The registration packet will only be viewed by the PI and co-investigator and will not be directly linked with any PHI to be created during the study. The Strider "Learn to Ride" intervention is designed to accommodate up to 10 children per intervention class, therefore no more than 10 participants will be recruited for the initial pilot study.

Outcome measures used will include the Pediatric Balance Scale (PBS), distance cycled, Participation and Environment Measure-Children and Youth (PEM-CY), and the PROMIS Physical Activity questionnaire. The PBS is a valid, 14-item assessment, developed based on the Berg Balance Scale. The PBS is a criterion-based measure, with each item scored on a 0-4 scale. Distance cycled will be measured based on the longest straight-line distance, out of three trials, that the participant is able to safely and independently propel their Strider bike. Previous research has used 100' as the distance criteria to identify mastery. The PEM-CY is participation level outcome measure used to assess a child's engagement in activities in the home, school, and community environments. The PEM-CY is a valid and reliable measure and is completed by parent/caregiver report, making it appropriate to use with children with DS. The parent/proxy PROMIS Physical Activity outcome measures assesses various aspects related to a child's participation in physical activity. Follow-up questionnaires (PEM-CY and PROMIS) will be sent by mail from the PI to the parent/caregiver to assess long-term changes in participation, time spent engaged in physical activity, and sustainability of the Strider bike intervention.

One the first day of the intervention, each participant will be assessed with the PBS to determine baseline balance ability. The initial straight-line distance, up to 100 feet, that each child can independently and safely ride their Strider balance bike will also be recorded. Additionally, each participants' parent/caregiver will be asked to complete the PEM-CY and the PROMIS questionnaire. This initial data collected will serve as each participants' baseline data. Each child will participate in five, consecutive, two-hour adaptive bike training sessions with instruction guided by the Strider "Learn to Ride" intervention. Each session will have no more than 10 participants. The biking sessions will be under the direct instruction of a pediatric physical therapist (the PI, Meredith Flowers) who has completed the certification to teach Strider "Learn to Ride" classes. Each session will take place in an indoor gym or paved, outdoor facility. Each participant will be fitted with an adaptive Strider bike to use for the duration of the 5-day intervention and to take home as their own, to encourage carry over, at the end of the training period. Each participant will also be required to provide and wear an appropriately fitted bike helmet when engaged in bike riding. Each session will begin with a 5-10-minute warm up, followed by at least 60 total minutes of riding activities based on the proven Strider "Learn to Ride" intervention. Individual participants will be allowed to take rest breaks as needed. Each session will conclude with 5-10 minutes of cool down activities. On the final day of the intervention, each participant will again be assessed with the PBS. The distance that each participant can safely and independently propel their Strider bike will be assessed and recorded. Each child's parent/caregiver will be contacted by mail from the PI to complete follow-up assessments at 3-, 6 months following completion of the initial intervention period. Outcome measures used for long-term follow up include the PEM-CY and PROMIS questionnaire. The PI and co-PI, both licensed physical therapists, will be assessing all participants.

IBM SPSS Statistics program will be used for all data analysis. Dependent t-tests will be used to analyze pre- and post-test scores of the PBS, PEM-CY, PROMIS and distance cycled. If the assumptions for the dependent t-test are not met, a Wilcoxon signed ranks test will be used to analyze the data.

ELIGIBILITY:
Inclusion Criteria:

* be between the ages of 5 and 17 years old with a diagnosis of Down syndrome
* have the core strength and balance necessary to maintain sitting on a two-wheel balance bike with their feet on the ground
* be able to follow simple commands.

Exclusion Criteria:

* significant cardiovascular event or illness in the past 6 months
* another medical diagnosis, besides Down syndrome, that would limit participation in the exercise programs.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meredith Flowers, DPT, Principal Investigator — University of Mississippi Medical Center, School of Physical Therapy
Locations (1):
- University of Mississippi Wellness Center, Flowood, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Balance Biking
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Balance Biking
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Pediatric Balance Scale (PBS) Mean Group Score
Description: The Pediatric Balance Scale (PBS) is a valid, 14-item assessment, developed based on the Berg Balance Scale, to assess balance in children. The PBS is a criterion-based measure, with each item scored on a 0-4 scale. The minimum score possible on the PBS is 0 points. The highest total score possible on the PBS is 56 points. Higher scores indicates better balance performance.The score reported is the mean PBS score of the group on day 5, the last day of the intervention.
Time Frame: Day 1 and Day 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Balance Biking
Number analyzed (Participants) | 7
score on a scale
  Pre-Intervention (Day 1) | 48.43 (4.467)
  Post-Intervention (Day 5) | 49.43 (3.552)
Statistical Analysis 1: Comparison: Balance Biking; Test type: Other — Wilcoxon signed ranks test used to compared pre-intervention to post-intervention means of the Pediatric Balance Scale. No power calculation performed or utilized; p < 0.05, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 1

2. Primary Outcome: Distance Biked
Description: How far, up to 100', that the child can independently ride their Strider bike
Time Frame: Day 1 and day 5
Population: Outcome of distance cycled assessed based on individual change scores (difference between distance cycled on day 1 and day 5). Group mean change scores also reported. No statistical analysis performed.
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | Balance Biking
Number analyzed (Participants) | 8
feet
  Pre-Intervention (Day 1) | 84 (30.69)
  Post-Intervention (Day 5) | 100 (0)

3. Primary Outcome: Change in Participation Level Based on the Participation and Environment Measure - Children and Youth (PEM-CY)
Description: The PEM-CY is participation level outcome measure used to assess a child's engagement in activities in the home, school, and community environments. The PEM-CY is a valid and reliable measure and is completed by parent/caregiver report, making it appropriate to use with children with DS. The PEM-CY asks questions related to 25 types of activiites that take place in the home, school, and community environments. Parents report "how often" their child has participated in each activity over the last 4 months (daily; few times a week; once a week; few times a month; once a month; few times in the last four months; once in the last four months; never); "how involved" their child is when participating in 1 or 2 activities that she or he does most often (5-very involved, 4, 3-somewhat involved, 2, 1-minimally involved); whether or not they want their child's participation to change and how they want it to change. The PEM-CY does not have scale scores or a total score.
Time Frame: 3 months, 6 months
Population: Data not reported due to not being collected secondary to participants submitting completed PEM-CYs.
Arm/Group | Balance Biking
Number analyzed (Participants) | 0

4. Primary Outcome: Change in Physical Activity Based on the Patient Reported Outcome Measure Information System (PROMIS) Physical Activity Measure - Proxy Report
Description: PROMIS Physical Activity outcome measures assesses various aspects related to a child's participation in physical activity.The PROMIS measure has 10 items that parents rate on a 5-point likert scale. A 1 indicates that the child participated in the activity "no days", 2 indicates that the child participated in the activity 1 day, 3 indicates that the child participated in the activity 2-3 days, 4 indicates that the child participated in the activity 4-5 days, and 5 indicates that the child participated in the activity 6-7 days. The PROMIS does not contain a total score.
Time Frame: 3 months, 6 months
Population: Data not reported due to participants not submitting completed PROMIS measure reports.
Arm/Group | Balance Biking
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Reported adverse events include events starting on day 0 and ending on day 5.
Arm/Group | Balance Biking
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-04): https://cdn.clinicaltrials.gov/large-docs/45/NCT03677245/Prot_SAP_000.pdf